CLINICAL TRIAL: NCT04724967
Title: Clinical Evaluation of CeraVe Hydrating Cleanser and Moisturizing Cream for the Improvement of Skin Condition in Patients With Diabetes Mellitus (DM) Related Skin Changes
Brief Title: CeraVe Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: CeraVe (Industry)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201149
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Complications
Keywords: cutaneous complication of DM
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CeraVe Group (Experimental): Participants in this group will receive the CeraVe Hydrating Cleanser and Moisturizing Cream for 28 days.
  Interventions: Drug: CeraVe Hydrating Cleanser; Drug: CeraVe Moisturizing Cream

INTERVENTIONS:
Drug: CeraVe Hydrating Cleanser — topical cleanser applied twice a day for 28 days
Drug: CeraVe Moisturizing Cream — topical cream applied twice a day for 28 days

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CeraVe Diabetic Skin Line for the improvement of skin condition in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 and 75 years of age.
2. Willing to provide written informed consent.
3. A diagnosis of diabetes mellitus (DM).
4. DM-related skin changes classified into one or more of the following four categories: i) skin lesions associated with DM; ii) infections; iii) cutaneous manifestations of DM complications; iv) skin reaction to DM treatment.

Exclusion Criteria:

1. History of allergy, anaphylaxis or hypersensitivity to any of the ingredients in CeraVe Hydrating Cleanser or Moisturizing Cream
2. History of allergic contact dermatitis secondary to cleansers or moisturizers.
3. Has a heightened immune response to common allergens, especially inhaled, topical or food allergens (atopy).
4. Has any clinical manifestation in the treatment are(s) or other disorders that, in the investigator's opinion, may affect assessments or the study products.
5. Inability to attend all study visits and follow treatment regimen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kirsner, MD/PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CeraVe Group
Started | 528
Completed | 528
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CeraVe Group
Number analyzed (Participants) | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327
  Male | 201
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes mellitus type [Count of Participants; unit: Participants]
  Type 1 | 92
  Type 2 | 436

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Adverse Events (AE)
Description: As evaluated by treating physician as possibly or probably related to intervention
Time Frame: Up to 33 days
Measure: Number; unit: percentage of participants
Arm/Group | CeraVe Group
Number analyzed (Participants) | 528
percentage of participants | 0

2. Primary Outcome: Percentage of Participants Reporting Adverse Events (AE)
Description: As evaluated by treating physician as possibly or probably related to intervention
Time Frame: Up to 33 days
Measure: Number; unit: percentage of participants
Arm/Group | CeraVe Group
Number analyzed (Participants) | 528
percentage of participants | 0

3. Primary Outcome: Number of Participants at Each GAIS Grading Scale
Description: Physician-assessed number of participants at each Global Aesthetic Improvement Scale (GAIS). GAIS has gradings of very much improved, much improved, improved, no change and worse. A grading of worse means the least aesthetic improvement.
Time Frame: At 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | CeraVe Group
Number analyzed (Participants) | 528
Participants
  Very much improved | 223
  Much improved | 224
  Improved | 72
  No change | 9
  Worse | 0

4. Primary Outcome: Number of Participants at Each Dry Skin Scale
Description: Physician-assessed number of participants at each Dry Skin Scale. Scales will be evaluated for each of the following conditions: roughness/scaling, itch, pain, erythema and fissures. Each condition will be scored from 0 (none), 1 (almost none), 2 (mild), 3 (moderate) to 4 (severe).
Time Frame: At 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | CeraVe Group
Number analyzed (Participants) | 528
Participants
  Roughness/scaling - none | 271
  Roughness/scaling - Almost None | 219
  Roughness/scaling - Mild | 28
  Roughness/scaling - Moderate | 7
  Roughness/scaling - Severe | 3
  Itchiness - None | 386
  Itchiness - Almost None | 116
  Itchiness - Mild | 21
  Itchiness - Moderate | 1
  Itchiness - Severe | 4
  Pain - None | 494
  Pain - Almost | 27
  Pain - Mild | 4
  Pain - Moderate | 1
  Pain - Severe | 2
  Erythema - None | 409
  Erythema - Almost None | 93
  Erythema - Mild | 19
  Erythema - Moderate | 6
  Erythema - Severe | 1
  Fissures - None | 408
  Fissures - Almost None | 104
  Fissures - Mild | 14
  Fissures - Moderate | 0
  Fissures - Severe | 2

ADVERSE EVENTS:
Time Frame: 33 days
Arm/Group | CeraVe Group
All-Cause Mortality (participants affected / at risk) | 0/528
Serious Adverse Events (participants affected / at risk) | 0/528
Other Adverse Events (participants affected / at risk) | 0/528

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT04724967/Prot_001.pdf